CLINICAL TRIAL: NCT06659887
Title: Effect of Different Low Flow Rates on Gas Exchange in Anesthetized Children During Apnea A Single Blinded Randomized Study
Brief Title: Different Low Flow Rates on Gas Exchange in Children During Apnea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yasser S Mostafa, MD (Other)
Responsible Party: Sponsor-Investigator, Yasser S Mostafa, MD, Lecturer of anesthesia, Fayoum University Hospital
Organization: Fayoum University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: D377
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Apnea
Keywords: Low flow rate; Children; Gas exchange
MeSH Terms: conditions — Apnea | interventions — Cannula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the clinically obvious oxygen administration modalities, study personnel in theatres cannot be blinded, but patients and parents will be blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low group (Active Comparator): Low flow 100% O2 AT 2 L/min
  Interventions: Device: nasal cannula
- Moderate group (Active Comparator): Low flow 100% O2 AT 4 L/min
  Interventions: Device: nasal cannula
- High group (Active Comparator): Low flow 100% O2 AT 8 L/min
  Interventions: Device: nasal cannula

INTERVENTIONS:
Device: nasal cannula — After induction, bag-mask ventilation with 100% oxygen and flow rates of 6 L/ min will be carried out until the expired oxygen concentration will be >90%, saturation of oxygen was 100%, and end tidal carbon dioxide was 30-40 mmHg. Once this will be reached, bag-mask ventilation will be stopped and apneic oxygenation will be initiated for 3 minutes
  Other Names: oxygen nasal cannula

SUMMARY:
Effect of Low flow apneic oxygenation in pediatrics on rate of accumulation of transcutaneous carbon dioxide also, had been studied, compared to high flow rates. Furthermore, a recent study in apneic anesthetized adult discussed the rate of accumulation of carbon dioxide in arterial blood during 4 min of apnea but, no study in pediatrics discussed the effect of different low flow rates on rate of carbon dioxide accumulation during a period of apnea.

Aim of the study: the authors aim to study the effect of different flow rates of low flow oxygenation during 3 min of apnea in anesthetized children on the rate of accumulation of carbon dioxide

DETAILED DESCRIPTION:
Introduction: During induction of general anesthesia using muscle relaxant, all patients experience a period of apnea which begins when mask ventilation is stopped prior to laryngoscopy and tracheal intubation and ends when ventilation is resumed. This period is a critical time as pediatrics especially infants and younger children are more liable for hypoxia than older children and adolescents. Hypoxia during this period of time in turn, had been proved to increase morbidity and mortality. Apneic oxygenation means uptake of oxygen by the blood from the lungs in the absence of spontaneous respiration or positive pressure ventilation, and its effectiveness in reducing the risk of hypoxemia during intubation in children had been proved. Many variables and outcomes had been studied during low flow apneic oxygenation in pediatrics and it was found that, it doesn't not only reduce the risk of hypoxemia but also prolongs of the safe apnea time up to 6 mins even when compared with high flow apneic oxygenation.

Anesthetic technique:

All children will undergo routine preoperative investigations: Complete blood count and coagulation profile. First, they will be examined as regards the fulfillment of inclusion criteria to be in the study or to be excluded from the study. Then, All children will receive premedication using midazolam 0.5 mg/kg intramuscular and intramuscular atropine 0.02 mg /kg.

Before induction of anaesthesia, patient characteristics and vital signs will be recorded {pulse oximetry, ECG, non-invasive blood pressure, end-tidal carbon dioxide}and will be applied all over the operation.

While establishing of IV access, all children will be preoxygenated using 6 liter/min of 100% O2 for 3 mins and if there will be a difficulty in obtaining an IV access, patients will be induced with inhaled sevoflurane followed by the placement of an IV cannula. Then, 2-3mg/Kg of Propofol, 1mcg/Kg of Fentanyl, and 0.3-0.5 mg/kg of Atracurium will be given. During induction of anesthesia an expert pediatric anesthesiologist will introduce an arterial radial cannula.

Intubation with an appropriate endotracheal will be started. After intubation a standardized manual airway recruitment maneuver will be performed. Mechanical ventilation will be started using pressure controlled-volume grantee mode and tidal volume will be adjusted to be 6 mg/kg/min and general anesthesia will be maintained using Isoflurane 1% minimum alveolar concentration. The lowest oxygen saturation and highest end-tidal carbon dioxide during the first five breaths will be recorded.

After recovery of all patients and before leaving the post anesthesia care unit(PACU), all parents will be asked about any postoperative side effects such as postoperative nausea and vomiting, stridor, coughing, laryngospasm, bronchospasm or pain.

Statistical analysis:

There is no published literature that covered the research idea to be used for sample sized calculation. So, we will conduct a pilot study of at least 5 patients in each group and use the obtained parameters for sample size calculation Statistical analysis will be performed using Statistical Package for the Social Sciences (SPSS) for Windows, version 29(IBM Corp., New York,USA). Descriptive statistics will be presented in the form of (mean ± SD), or (median and interquartile range) for numerical data, while numbers and percentages will be used for categorical data.

Testing for normality of distribution will be done using the Shapiro-Wilk test. Categorical variables will be analyzed using Chi-square test or Fisher's exact test. Differences in parametric normally distributed data will be compared using Student's t-tests, while the non-parametric data will be compared using Mann-Whitney U-test. Results will be considered statistically significant if P value is less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 6 years old weighting 10-20 kg.
* American Society of Anesthesiologists (ASA) physical status I or II.
* Children will be scheduled for elective surgery under general anesthesia.

Exclusion Criteria:

* Parent refusal
* Patient required nasal intubation
* Children with a cardio-respiratory disease like asthma or recent upper respiratory infection.
* Anemia.
* Obstructive sleep apnea, sepsis.
* Children prone to hypoxia or hypercarbia, and upper airway obstruction.
* Children reported to have nasal obstruction .

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
rise of arterial pressure of carbon dioxide | between 60s and 180s time points of apnea
  mmHg

SECONDARY OUTCOMES:
Time to oxygen desaturation | 5 seconds after the onset of apnea
  below 95%
Number of patients reached 6 minutes of apnea | 1 minute after end of apneic oxygenation
  Count number of patients in each group
Pressure difference between the end-tidal carbon dioxide and the arterial carbon dioxide | Between the end of apnea and the preceding blood gas
  mmHg
Mean difference in arterial pressure of oxygen | at the beginning of apnea
  mmHg
Mean difference in arterial pressure of oxygen | at the end of apnea time
  mmHg
Lowest recorded oxygen saturation | throughout the apneic oxygenation
  in percentage (%)
Heart rate | Before anaesthetizing child
  beat/minute
Mean arterial blood pressure | Before anaesthetizing child
  mmHg
Heart rate | During apnea time
  beat/minute
Mean arterial blood pressure | During apnea time
  mmHg
Occurence of sore throat | in first postoperative day
  Yes or no

OTHER OUTCOMES:
Age | 1 hour preoperatively
  Years
Weight | 1 hour preoperatively
  Kilogram

CONTACTS AND LOCATIONS:
Overall Officials: Safaa G Ragab, MD, Study Director — Fayoum University; Ahmed A Lotfy, MD, Study Director — Fayoum University
Locations (1):
- Fayoum University Hospital, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li S, Hsieh TC, Rehder KJ, Nett S, Kamat P, Napolitano N, Turner DA, Adu-Darko M, Jarvis JD, Krawiec C, Derbyshire AT, Meyer K, Giuliano JS Jr, Tala J, Tarquinio K, Ruppe MD, Sanders RC Jr, Pinto M, Howell JD, Parker MM, Nuthall G, Shepherd M, Emeriaud G, Nagai Y, Saito O, Lee JH, Simon DW, Orioles A, Walson K, Vanderford P, Shenoi A, Lee A, Bird GL, Miksa M, Graciano AL, Bain J, Skippen PW, Polikoff LA, Nadkarni V, Nishisaki A; for National Emergency Airway Registry for Children (NEAR4KIDS) and Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Frequency of Desaturation and Association With Hemodynamic Adverse Events During Tracheal Intubations in PICUs. Pediatr Crit Care Med. 2018 Jan;19(1):e41-e50. doi: 10.1097/PCC.0000000000001384. PMID 29210925
- [Background] Parker MM, Nuthall G, Brown C 3rd, Biagas K, Napolitano N, Polikoff LA, Simon D, Miksa M, Gradidge E, Lee JH, Krishna AS, Tellez D, Bird GL, Rehder KJ, Turner DA, Adu-Darko M, Nett ST, Derbyshire AT, Meyer K, Giuliano J Jr, Owen EB, Sullivan JE, Tarquinio K, Kamat P, Sanders RC Jr, Pinto M, Bysani GK, Emeriaud G, Nagai Y, McCarthy MA, Walson KH, Vanderford P, Lee A, Bain J, Skippen P, Breuer R, Tallent S, Nadkarni V, Nishisaki A; Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Relationship Between Adverse Tracheal Intubation Associated Events and PICU Outcomes. Pediatr Crit Care Med. 2017 Apr;18(4):310-318. doi: 10.1097/PCC.0000000000001074. PMID 28198754
- [Background] Dias R, Dave N, Chhabria R, Shah H, Garasia M. A randomised comparative study of Miller laryngoscope blade versus Oxiport(R) Miller laryngoscope blade for neonatal and infant intubations. Indian J Anaesth. 2017 May;61(5):404-409. doi: 10.4103/ija.IJA_86_17. PMID 28584350